CLINICAL TRIAL: NCT06551064
Title: A Randomized, Double-Blind, Multicenter, Pharmacokinetic Equivalence Clinical Trial of Adjuvant FYB206 (Keytruda Biosimilar Candidate) in Comparison With Keytruda (Pembrolizumab) to Demonstrate Pharmacokinetic Similarity in Patients With Completely Resected Stage IIB/IIC or Stage III Melanoma
Brief Title: Assessment of PK Similarity of FYB206 in Comparison With Keytruda in Resected Stage II or III Melanoma Patients
Acronym: Dahlia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Formycon AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FYB206-C1-01; 2023-509765-20-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Melanoma, Stage II; Melanoma Stage III
Keywords: pembrolizumab; biosimilar; melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- FYB206 (Experimental)
  Interventions: Biological: FYB206
- Keytruda (Active Comparator)
  Interventions: Biological: Keytruda

INTERVENTIONS:
Biological: FYB206 — FYB206 (Keytruda biosimilar candidate - test product) 200 mg administered as an IV infusion over 30 minutes on Day 1 of each cycle
  Arms: FYB206
Biological: Keytruda — Keytruda (reference product) 200 mg administered as an IV infusion over 30 minutes on Day 1 of each cycle
  Arms: Keytruda

SUMMARY:
Melanoma is a kind of skin cancer that starts in the melanocytes. Melanocytes are cells that make the pigment that gives skin its colour. 'Resected' means the melanoma has been completely removed with surgery.

Pembrolizumab is an anti-cancer therapy that works with the immune system to fight cancer cells. Some cancer cells develop a way to hide from the body's immune system and, thus, allow the cancer cells to spread and grow. Pembrolizumab helps the immune system recognize and kill these cancer cells that want to hide.

Pembrolizumab is a biologic drug (produced by living organisms) available in the market under the brand name Keytruda. Keytruda is approved globally for the treatment of a variety of cancers and as an addon or after therapy to primary cancer treatment like surgery. This helps prevent the cancer from returning, improving overall survival.

FYB206 is a proposed biosimilar to Keytruda. A biosimilar is not identical but very similar to its original biologic. Biosimilars are expected to have a similar effect and safety to the original biologic. To learn what happens to a drug once it is in the body is called pharmacokinetics (PK). PK for biosimilar drugs is expected to remain similar to the original biologic. This study is to show that PK of FYB206 is similar to the reference product Keytruda for patients with completely resected Stage IIB/IIC or Stage III melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage IIB, IIC, or III histologically confirmed cutaneous melanoma (as classified by the American Joint Committee on Cancer [AJCC]'s Cancer Staging Manual, 8th Edition) who have undergone complete resection within 12 weeks before randomization. No evidence of past or current satellites or in-transit metastases.
* Disease status for the post-surgery baseline assessment must be documented by full chest/abdomen/pelvis computed tomography (CT) and/or magnetic resonance imaging (MRI) with neck CT and/or MRI (for head and neck primaries) and must have completed a clinical examination after the informed consent form has been signed and before enrollment.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
* Caucasian adult patients ≥18 years of age on the day of signing the informed consent.

Exclusion Criteria:

* History of radiation therapy for melanoma before trial entry. Post-lymph node dissection radiotherapy is allowed; however, this should be completed at least 7 days before treatment starts.
* Uveal or ocular melanoma.
* Diagnosis of immunodeficiency or receiving long-term systemic steroid therapy (>10 mg/day of prednisone or equivalent) or any other form of immunosuppressive therapy ≤7 days before the first dose of IMP.
* Received prior therapy with an anti-cytotoxic T-lymphocyte antigen-4 (CTLA-4) monoclonal antibody (eg, ipilimumab), anti-programmed cell death 1 (PD-1), anti-programmed cell death ligand 1 (PD-L1), or anti-programmed cell death ligand 2 (PD-L2) agent or agent directed to another stimulatory or co-inhibitory T-cell receptor.
* Received prior systemic anticancer therapy for melanoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
AUCtau,sd at Cycle 1 | 21 days
  Area under the concentration curve for one dosing interval (tau=21 days) after a single (initial) dose (AUCtau,sd) of FYB206 and Keytruda (Cycle 1)
AUCtau,sd at Cycle 6 | 126 days
  Area under the concentration curve for one dosing interval (tau=21 days) at steady state (AUCtau,ss) of FYB206 and Keytruda (Cycle 6)

CONTACTS AND LOCATIONS:
Locations (17):
- Formycon Investigative Site, Sarajevo, Bosnia and Herzegovina
- Formycon Investigative Site, Sofia, Bulgaria
- Formycon Investigative Site, Tartu, Estonia
- Georgia (3):
  - Formycon Investigative Site, Batumi
  - Formycon Investigative Site, Kutaisi
  - Formycon Investigative Site, Tbilisi
- Formycon Investigative Site, Kaunas, Lithuania
- Formycon Investigative Site, Chisinau, Moldova
- Formycon Investigative Site, Skopje, North Macedonia
- Poland (2):
  - Formycon Investigative Site, Krakow
  - Formycon Investigative Site, Lodz
- Romania (2):
  - Formycon Investigative Site, Bucharest
  - Formycon Investigative Site, Cluj-Napoca
- Serbia (3):
  - Formycon Investigative Site, Belgrade
  - Formycon Investigative Site, Kragujevac
  - Formycon Investigative Site, Niš
- Formycon Investigative Site, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No